CLINICAL TRIAL: NCT04087668
Title: Deep Sedation and General Anesthesia for Endoscopic Retrograde Cholangiopancreatography
Brief Title: Different Anesthetic Technique For ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-SR-205
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia; Adverse Effect
Keywords: ERCP; General anesthesia; Endoscopy; MAC
MeSH Terms: interventions — Anesthesia, General; Neoadjuvant Therapy; Neuromuscular Blockade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monitored Anesthesia Care (Other): Patients in this arm will undergo an ERCP using monitored anesthesia care (MAC) with propofol based deep sedation.
  Interventions: Procedure: Monitored Anesthesia Care
- General Anesthesia (Other): Patients in this arm will receive standard general anesthesia with neuromuscular blockade.
  Interventions: Procedure: General Anesthesia
- General Anesthesia Without Neuromuscular Blockade (Other): Patients in this arm will receive nasotracheal intubation without neuromuscular blockade.
  Interventions: Procedure: Induction Without Neuromuscular Blockade

INTERVENTIONS:
Procedure: Monitored Anesthesia Care — MAC was induced and maintained via the continuous infusion of propofol AND remifentanil using a target-controlled infusion (TCI) pump. The appropriate level of sedation was 65 to 80 points on BIS. The adjunctive sedatives (eg, fentanyl, midazolam) was at the discretion of the anesthesia team.
  Arms: Monitored Anesthesia Care
Procedure: General Anesthesia — Induction was done with propofol (2 mg/kg) , cis-atracurium (0.15 mg/kg) , and fentanyl (5μg/kg). After orotracheal intubation, general anesthesia was maintained with sevoflurane (1-1.3MAC) , propofol (3mg/kg/h), remifentanil (0.05-0.2 ug/kg/min) and repetitive doses of 0.1mg atracurium per kilogram were administered. After the procedure was completed, neostigmine mixed with atropine was used as a reversal agent for the neuromuscular blockade, and the patient was extubated when the recovery from anesthesia was confirmed.The BIS was 45 to 60 points .
  Arms: General Anesthesia
Procedure: Induction Without Neuromuscular Blockade — Anaesthesia was induced with propofol (2 mg/kg), remifentanil(3 ug/kg) and 2% lidocaine (1 mg/kg). Nasotracheal intubation was performed 60 s after the administration. After intubation, general anesthesia was sevoflurane (1-1.3MAC) , propofol (3mg/kg/h), remifentanil (0.05-0.2 ug/kg/min). After the procedure was completed, the patient was extubated when the recovery from anesthesia was confirmed.The BIS was 45 to 60 points .
  Arms: General Anesthesia Without Neuromuscular Blockade

SUMMARY:
Providing the appropriate anesthetic technique for endoscopic retrograde cholangiopancreatography (ERCP) in remote locations can be challenging. The aim of this study was therefore to prospectively assess and compare the feasibility of monitored anesthesia care (MAC) with propofol based deep sedation, standard general anesthesia and general anesthesia without neuromuscular blockade in patients undergoing ERCP.

DETAILED DESCRIPTION:
ERCP is identified as one of the most invasive endoscopic procedures, during which patients may experience anxiety, discomfort and suffer different degree of pain. So, anesthesia and analgesia are essential for this invasive procedure, especially therapeutic ERCPs. Thus, we compared the efficacy of using monitored anesthesia care (MAC) with deep sedation versus general anesthesia (GA) to perform this procedure and the incidence of complications associated with these methods of anesthesia.

Previous studies have concluded that intubation is possible without the use of neuromuscular blockade. We assume that the use of propofol and adjuvants short-acting opioids may provide adequate conditions for tracheal intubation. It was also hypothesized that it may also be useful in facilitating ERCP under general anesthesia without neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years old
* Grade Ⅰ and Ⅲ according to physical status classification system of the American Society of Anesthesiologists (ASA)
* Coagulation function tests in normal range

Exclusion Criteria:

* Potentially difficult airways
* Administration of sedative or narcotic drugs in the previous 24 hours
* Severe renal or hepatic impairment
* Severe cardiopulmonary comorbidities (defined as American Society of Anesthesiologists physical status IV or greater)
* Contraindications to a nasotracheal intubation
* Coagulopathy
* History of frequent episodes of epistaxis
* Emergent ERCP
* At risk for reflux and aspiration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The overall complication rate | within 72 hours of ERCP
  The primary outcome was the overall pulmonary and cardiac complication rate.

SECONDARY OUTCOMES:
Conversion to GA | During the procedure
  Conversion to general anesthesia
Temporary interruption rate of ERCP | During the procedure
Premature termination rate of ERCP | During the procedure
Procedural failure rate of ERCP | During the procedure
Procedure time | During the procedure
Anesthesia time | During the procedure
Room time | During the procedure
  Patient room-in to room-out time in the ERCP suite ("room time").
Immediate Adverse Events | within 24 hours of ERCP
Delayed Adverse Events | within 72 hours of ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Cao, Study Chair — The First Affiliated Hospital with Nanjing Medical University; Junbei Wu, Study Director — The First Affiliated Hospital with Nanjing Medical University; Nana Li, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Xiaoyang Tang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Jigang Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith A, Silvestro L, Rodriguez RE, Austin PN. Evidence-Based Selection of Sedation Agents for Patients Undergoing Endoscopic Retrograde Cholangiopancreatography. Gastroenterol Nurs. 2016 Jan-Feb;39(1):32-41. doi: 10.1097/SGA.0000000000000195. PMID 26825562
- [Background] Yang JF, Farooq P, Zwilling K, Patel D, Siddiqui AA. Efficacy and Safety of Propofol-Mediated Sedation for Outpatient Endoscopic Retrograde Cholangiopancreatography (ERCP). Dig Dis Sci. 2016 Jun;61(6):1686-91. doi: 10.1007/s10620-016-4043-3. Epub 2016 Jan 29. PMID 26825844
- [Background] Barnett SR, Berzin T, Sanaka S, Pleskow D, Sawhney M, Chuttani R. Deep sedation without intubation for ERCP is appropriate in healthier, non-obese patients. Dig Dis Sci. 2013 Nov;58(11):3287-92. doi: 10.1007/s10620-013-2783-x. Epub 2013 Jul 23. PMID 23877477
- [Background] Coghlan SF, McDonald PF, Csepregi G. Use of alfentanil with propofol for nasotracheal intubation without neuromuscular block. Br J Anaesth. 1993 Jan;70(1):89-91. doi: 10.1093/bja/70.1.89. PMID 8431342
- [Background] Grant S, Noble S, Woods A, Murdoch J, Davidson A. Assessment of intubating conditions in adults after induction with propofol and varying doses of remifentanil. Br J Anaesth. 1998 Oct;81(4):540-3. doi: 10.1093/bja/81.4.540. PMID 9924229
- [Background] Erhan E, Ugur G, Gunusen I, Alper I, Ozyar B. Propofol - not thiopental or etomidate - with remifentanil provides adequate intubating conditions in the absence of neuromuscular blockade. Can J Anaesth. 2003 Feb;50(2):108-15. doi: 10.1007/BF03017840. PMID 12560298
- [Background] Klemola UM, Mennander S, Saarnivaara L. Tracheal intubation without the use of muscle relaxants: remifentanil or alfentanil in combination with propofol. Acta Anaesthesiol Scand. 2000 Apr;44(4):465-9. doi: 10.1034/j.1399-6576.2000.440419.x. PMID 10757583